CLINICAL TRIAL: NCT04419558
Title: Zephyrus II: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Efficacy and Safety Study of Pamrevlumab in Subjects With Idiopathic Pulmonary Fibrosis (IPF)
Brief Title: Zephyrus II: Efficacy and Safety Study of Pamrevlumab in Participants With Idiopathic Pulmonary Fibrosis (IPF)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Kyntra Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FGCL-3019-095
Record Dates: First submitted 2020-06-03; First posted 2020-06-05 (Actual); Results first posted 2024-08-12 (Actual); Last update posted 2024-08-12 (Actual); Status verified 2024-08

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; IPF; Idiopathic Interstitial Pneumonia; Interstitial Lung Disease; Lung Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis; Idiopathic Interstitial Pneumonias; Lung Diseases, Interstitial; Pulmonary Fibrosis | interventions — pamrevlumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: During the Open-label extension phase, all participants will receive pamrevlumab in an open-label manner. No unblinding of participant's treatment assignment in the treatment phase (main study) will occur for purposes of open-label extension participation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pamrevlumab (Experimental): Treatment phase: Pamrevlumab 30 mg/kg administered by IV infusion, every 3 weeks, for a total of up to 17 infusions over 48 weeks.
  Open-label extension phase: Pamrevlumab 30 mg/kg administered by intravenous infusion, every 3 weeks for up to 48 weeks
  Interventions: Drug: Pamrevlumab
- Placebo (Experimental): Pamrevlumab-matching placebo administered by IV infusion every 3 weeks for a total of up to 17 infusions over 48 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pamrevlumab — Sterile solution for injection
  Other Names: FG-3019
  Arms: Pamrevlumab
Drug: Placebo — Sterile solution for injection
  Arms: Placebo

SUMMARY:
This is a Phase 3 trial to evaluate the efficacy and safety of 30 milligrams (mg)/kilogram (kg) intravenous (IV) infusions of pamrevlumab administered every 3 weeks as compared to placebo in participants with Idiopathic Pulmonary Fibrosis (IPF). There is a 48-week randomized treatment phase followed by an optional, open-label extension phase.

DETAILED DESCRIPTION:
The intent of this study is to evaluate the efficacy and safety of pamrevlumab as monotherapy in participants with IPF. Participants who are not being treated with approved IPF therapies (that is, nintedanib or pirfenidone) may be eligible for screening. Examples of reasons participants may not be treated with approved IPF therapies include but are not limited to:

* Intolerant or not responsive to approved IPF therapies
* Ineligible to receive these therapies
* Participant voluntarily declines to receive approved IPF therapies after being fully informed of the potential benefits/risks

NOTE: No participant should discontinue an approved IPF therapy for the purpose of enrolling in this study.

During the 48-week treatment phase of the study, co-administration of an approved IPF therapy (such as, pirfenidone or nintedanib) is acceptable if clinically indicated in the Investigator's opinion, after assessment of potential risks/benefits of such combination with blinded study treatment.

Participants who complete the 48-week study will be eligible for an optional, open-label extension phase with continued access to pamrevlumab, regardless of their randomized assignment.

ELIGIBILITY:
Key Inclusion Criteria:

1. Diagnosis of IPF as defined by American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Latin American Thoracic Association (ATS/ERS/JRS/ALAT) guidelines within the past 7 years prior to study participation.
2. High-resolution computed tomography (HRCT) scan at Screening, with ≥10% to <50% parenchymal fibrosis (reticulation) and <25% honeycombing.
3. FVCpp value >45% and <95% at Screening and Day 1 (prior to randomization).
4. Diffusing capacity of the lungs for carbon monoxide (DLCO) percent predicted ≥25% and ≤90%.
5. Not currently receiving treatment for IPF with an approved therapy for IPF (such as, pirfenidone or nintedanib) for any reason, including prior intolerance or lack of response to an approved IPF therapy, or choice to forego treatment with an approved IPF therapy after a full discussion with the Investigator regarding risks/benefits of such therapy.

Key Exclusion Criteria:

1. Previous exposure to pamrevlumab.
2. Evidence of significant obstructive lung disease, as evidenced by spirometry or HRCT.
3. Female participants who are pregnant or nursing.
4. Smoking within 3 months of Screening and/or unwilling to avoid smoking throughout the study.
5. Interstitial lung disease other than IPF.
6. Sustained improvement in the severity of IPF during the 12 months prior to screening.
7. Other types of respiratory diseases that, in the opinion of the Investigator, would impact the primary protocol endpoint or otherwise preclude participation in the study, including diseases of the airways, lung parenchyma, pleural space, mediastinum, diaphragm, or chest wall.
8. Certain medical conditions, that, in the opinion of the Investigator, would impact the primary protocol endpoint or otherwise preclude participation in the study (such as, myocardial infarction/stroke, severe chronic heart failure, pulmonary hypertension, or cancers).
9. Acute IPF exacerbation during Screening or Randomization including hospitalization due to acute IPF exacerbation within 4 weeks prior to or during screening.
10. Use of any investigational drugs or unapproved therapies, or participation in any clinical trial with an investigational new drug within 30 days prior to screening. Or use of approved IPF therapies (such as, pirfenidone or nintedanib) within 1 week prior to screening.
11. History of allergic or anaphylactic reaction to human, humanized, chimeric or murine monoclonal antibodies, or to any component of the excipient.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2020-09-30 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (157):
- United States (23):
  - UAB Lung Health Center, Birmingham, Alabama
  - UC San Francisco, San Francisco, California
  - National Jewish Health, Denver, Colorado
  - Yale University, New Haven, Connecticut
  - St. Francis Medical Center, Clearwater, Florida
  - Pulmonary Disease Specialists d/b/a PDS Research, Kissimmee, Florida
  - TGH/USF Center for Advanced Lung Disease and Lung Transplant, Tampa, Florida
  - Emory University/The Emory Clinic, Atlanta, Georgia
  - University of Iowa, Iowa City, Iowa
  - The University of Kansas Medical Center, Kansas City, Kansas
  - University of Maryland Medical Center, Baltimore, Maryland
  - The General Hospital Corporation d/b/a Massachusetts General Hospital, Boston, Massachusetts
  - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Duke University Medical Center, Durham, North Carolina
  - PulmonIx, LLC, Greensboro, North Carolina
  - Ohio State University, Columbus, Ohio
  - Penn State Milton S Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Low Country Lung and Critical Care, PA, Charleston, South Carolina
  - The University of Vermont, Burlington, Vermont
  - University of Wisconsin Clinical Research, Madison, Wisconsin
- Fundacion Respirar - Centro Médico Dra. De Salvo, Ciudad Autonoma de Buenos Aires (caba), Argentina
- Brazil (9):
  - Hospital das Clínicas da UFMG - Centro de Pesquisas Clínicas do Hospital das Clínicas da Universidade Federal de Minas Gerais - CPC HC/UFMG, Belo Horizonte, Minas Gerais
  - Irmandade da Santa Casa de Misericórdia de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - HSL-PUCRS Hospital São Lucas da Pontifícia Universidade Católica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - Hospital Dia do Pulmão, Blumenau, Santa Catarina
  - Unidade de Pesquisa Clínica da Faculdade de Medicina de Botucatu - UPECLIN - UNESP, Botucatu, São Paulo
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos LTDA EPP, São Bernardo do Campo, São Paulo
  - CPQuali Pesquisa Clínica Ltda., São Paulo
  - Hospital Alemao Oswaldo Cruz, São Paulo
  - INCOR - Instituto do Coração Centro de Pesquisa Prof. Dr. Fulvio Pileggi Hospital das Clínicas da Faculdade de Medicina da USP - HCFMUSP, São Paulo
- China (15):
  - BeiJing Chao-Yang Hospital,Capital Medical University, Beijing
  - Beijing Frindship hosiptal capital Medical University, Beijing
  - China Japan Friendship hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - Sichuan People's Hospital, Chengdu
  - Guangdong Provincial People's Hospital, Guangzhou
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou
  - Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Oriental Hospital, Shanghai
  - The First Hospital of China Medical University, Shenyang
  - General Hospital of Tianjin Medical University, Tianjing
  - Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - The Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an
  - General Hospital of Ningxia Medical University, Yinchuan
- Colombia (3):
  - Fundación Santa Fe de Bogotá, Bogotá
  - Fundación Neumológica Colombiana, Bogotá
  - Healthy Medical Center S.A.S, Zipaquirá
- Czechia (3):
  - Fakultní nemocnice Brno, Brno
  - Nemocnice Jihlava, Jihlava
  - Nemocnice Na Bulovce, Klinika pneumologie, Prague
- Denmark (2):
  - Aarhus Universitets Hospital, Aarhus
  - Odense University Hospital, Odense
- Dominican Republic (2):
  - Centro de Obstetricia y Ginecologia, Santo Domingo
  - Centro Medico Dominicano, Santo Domingo
- France (10):
  - University Hospital Avicenne, Bobigny
  - Hôpital Cardio-Vasculaire et Pneumologique Louis Pradel, Bron
  - CHU de Caen, Caen
  - Centre Memoire Ressources Recherche, Hopital F. MITTERRAND, Dijon
  - C.H.R.U. de Montpellier - Hôpital Lapeyronie, Montpellier
  - CHU de Nice Hôpital Pasteur, Nice
  - Hôpital Bichat - Claude Bernard, Paris
  - CHU de Reims Hopital Maison Blanche, Reims
  - CHU de Rennes Hôpital Pontchaillou, Rennes
  - Service de Néphrologie, Hôpital Bretonneau, CHRU de Tours, Tours
- Georgia (2):
  - Research Institute Of Clinical Medicine Todua Clinic, Tbilisi
  - Clinic Diacor, Tbilisi
- Germany (7):
  - Ruhrlandklinik-Universitaetsmedizin Essen, Essen
  - Klinik Schillerhoehe, Gerlingen
  - Agaplesion Evangelisches Krankenhaus Mittelhessen, Giessen
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - University of Munich, Munich
  - RoMed Klinikum Rosenheim, Rosenheim
  - Institut fur Pneumologie an der Universitat zu Koln, Solingen
- Hungary (4):
  - Semmelweis University Clinic of Pulmonology, Budapest
  - Orszagos Koranyi Tbc es Pulmonologiai Intezet, IV. Tudobelosztaly, Budapest
  - Fejer Megyei Szent Gyorgy kh, Székesfehérvár
  - Pulmonology Hospital, Törökbálint
- Royal College of Surgeons in Ireland, Dublin, Ireland
- Italy (11):
  - Gaspare Rodiloco Hospital, Catania
  - Ospedale G.B.Morgagni L.Pierantoni - Azienda Unita Sanitaria Locale (AUSL) di Forli, Forlì
  - Ospedale San Giuseppe, Milan
  - AOU Policlinico di Modena, Modena
  - Monaldi Hospital, Naples
  - Azienda Ospedaliera Universitaria di Padova, Padua
  - IRCCS Fondazione San Matteo di Pavia, Pavia
  - Agostina Gemelli University Polyclinic, Rome
  - Azienda Ospedaliera Universitaria Senese, Policlinico "Le Scotte", Siena
  - Azienda Ospedaliera Citta' della Salute e delle Scienza di Torino, Torino
  - Azienda Ospedaliero-Universitaria "Ospedali Riuniti di Ancona", Torrette
- Lebanon (3):
  - American University of beirut medical center, Beirut
  - Hotel Dieu De France, Beirut
  - Rafik Hariri University Hospital (Clinical Research Unit), Bir Hassan
- Mexico (6):
  - Instituto Nacional de Enfermedades Respiratorias INER, México
  - Unidad Medica para la Salud Integral (UMSI), México
  - Medical Care and Research S.A. de C.V., México
  - St. Lucas Clinical Research Center SA de CV, México
  - Centro Regional para el estudio del Adulto Mayor, Servicio de Geriatria, Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Oaxaca Site Management Organization S.C. (OSMO), Oaxaca City
- Netherlands (5):
  - Dept. of Pulmonary Diseases, Amsterdam
  - Catharina Hospital, Eindhoven
  - Longarts - Opleider Longziekten Zuyderland MC, Heerlen
  - St. Antonius Ziekenhuis BV, Nieuwegein
  - Canisius-Wilhelmina Ziekenhuis, Nieuwegein
- Peru (6):
  - Clinica Internacional, Lima
  - Clinica San Pablo, Lima
  - Clinica Providencia, Lima
  - Hospital Nacional Cayetano Heredia / Servicio de Inmunología y Reumatología, Lima
  - Centro de Investigacion Ricardo Palma, San Isidro
  - Clinica La luz, Santa Beatriz
- Poland (5):
  - Centrum Dentystyczno-Lekarskie Promedica Joanna Markiewicz, Będzin
  - Centrum Medycyny Oddechowej Mroz SJ, Bialystok
  - Gornoslaskie Centrum Medyczne im. prof. Leszka Gieca Slaskiego Uniwersytetu Medycznego w Katowicach, Katowice
  - University Hospital No1, Lodz
  - Instytut Gruzlicy i Chorob Pluc, Warsaw
- Serbia (4):
  - Municipal Institute for Lung Diseases and Tuberculosis, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Diseases of Vojvodina, Kamenitz
  - University Clinical Center of Nis, Niš
- South Korea (15):
  - Myongji Hospital, Goyang-si, Gyeonggi-do
  - Soonchunhyang University Hospital Bucheon, Bucheon-si
  - The Catholic University of Korea Bucheon St. Mary's Hospital, Bucheon-si
  - Inje University Haeundae Paik Hospital, Busan
  - Inje University Hospital Iisan Paik Hospital, Goyang
  - Chonnam National University Hospital, Gwangju
  - Gachon University Gil Medical Centre, Incheon
  - Seoul National University Bundang Hospital, Seongnam
  - Seoul National University Hospital, Seoul
  - Kyunghee University Medical Center, Seoul
  - Severance hospital, Seoul
  - Soonchunhyang University Hospital Seoul, Seoul
  - Asan Medical Center, Seoul
  - The Catholic University of Korea, Yeouido ST. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (8):
  - Hospital Universitario de Bellvitge, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitaio de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Clinico San Carlos-Madrid C/Martin Lagos s/n, Madrid
  - Hospital Universitario Quironsalud Madrid, Madrid
  - Hospital Universitario Marques de Valdecilla, Santander
  - Hospital Universitario Nuestra Senora de Valme, Seville
- Universitätsklinik für Pneumologie, Bern, Switzerland
- Ukraine (3):
  - Communal non-profit enterprise "City clinical hospital #16" of Dnipro Сit Сouncil, Dnipro
  - Ivano-Frankivsk Regional Phthisiology-Pulmonology Center of Ivano-Frankivsk regional council, Ivano-Frankivsk
  - National Institute of Phthisiology and Pulmonology named after F. G. Yanovskyi NAMS of Ukraine, Clinical and Functional Department, Kyiv
- United Kingdom (8):
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Queen Elizabeth Hospital, University Hospitals Birmingham NHS Foundation Trust, Birmingham
  - Papworth Hospital NHS Foundation Trust, Advanced Heart Failure Unit, Cambridge
  - The Princess Alexandra Hospital NHS Trust, Harlow
  - Royal Brompton Hospital, London
  - University College London, London
  - Manchester University NHS Foundation Trust, Manchester
  - Southampton General Hospital, Southampton

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study included a Double-blind (DB) Period and an Open-label Extension (OLE) Period.
Groups:
- Pamrevlumab: Participants received pamrevlumab 30 milligrams (mg)/kilogram (kg), administered by intravenous (IV) infusion, every 3 weeks, for a total of up to 17 infusions over 48 weeks in the DB period. Participants who completed the treatment in DB period and entered in the OLE period, continued to receive pamrevlumab 30 mg/kg administered by IV infusion, every 3 weeks for up to 48 weeks.
- Placebo: Participants received pamrevlumab-matching placebo, administered by IV infusion every 3 weeks for a total of up to 17 infusions over 48 weeks in the DB period. Participants who completed the treatment in DB period and entered in the OLE period, received pamrevlumab 30 mg/kg administered by IV infusion, every 3 weeks for up to 48 weeks.
Period: DB Period (48 Weeks)
Arm/Group | Pamrevlumab | Placebo
Started | 184 | 188
Received at Least 1 Dose of Study Drug | 183 | 188
Completed | 47 | 56
Not Completed | 137 | 132
Not completed — Adverse Event | 6 | 6
Not completed — Death | 14 | 11
Not completed — Lost to Follow-up | 1 | 3
Not completed — Investigator Decision | 0 | 1
Not completed — Study terminated by sponsor | 99 | 101
Not completed — Disease Progression | 1 | 0
Not completed — Withdrawal by Subject | 11 | 7
Not completed — Lung Transplant | 1 | 0
Not completed — Participant Decision | 4 | 3
Period: OLE Period (48 Weeks)
Arm/Group | Pamrevlumab | Placebo
Started | 41 | 45
Completed | 0 | 0
Not Completed | 41 | 45
Not completed — Adverse Event | 3 | 1
Not completed — Death | 4 | 6
Not completed — Study terminated by sponsor | 34 | 37
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all randomized participants.
Groups:
- Pamrevlumab: Participants received pamrevlumab 30 mg/kg, administered by IV infusion, every 3 weeks, for a total of up to 17 infusions over 48 weeks in the DB period. Participants who completed the treatment in DB period and entered in the OLE period, continued to receive pamrevlumab 30 mg/kg administered by IV infusion, every 3 weeks for up to 48 weeks.
- Total: Total of all reporting groups
Arm/Group | Pamrevlumab | Placebo | Total
Number analyzed (Participants) | 184 | 188 | 372
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.2 (7.8) | 70.1 (8.2) | 70.1 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 44 | 89
  Male | 139 | 144 | 283
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 52 | 45 | 97
  Not Hispanic or Latino | 125 | 141 | 266
  Unknown or Not Reported | 7 | 2 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 42 | 55 | 97
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 111 | 114 | 225
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 29 | 16 | 45
Forced Vital Capacity (FVC) [Mean (Standard Deviation); unit: liters] — FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Population: 'Number analyzed' = participants evaluable for this baseline measure.
  liters
    number analyzed (Participants) | 184 | 187 | 371
    (all) | 2.4811 (0.6477) | 2.5097 (0.6573) | 2.4955 (0.6518)

OUTCOME MEASURES:

1. Primary Outcome: DB Period: Change From Baseline in FVC at Week 48
Description: FVC is a standard pulmonary function test used to quantify respiratory muscle weakness. FVC was the volume of air that can forcibly be blown out after full inspiration in the upright position, measured in liters. Least square (LS) mean and standard error (SE) were analyzed using mixed model repeated measures (MMRM).
Time Frame: Baseline, Week 48
Population: The ITT population included all randomized participants. Here, 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 70 | 76
liters | -0.30 (0.057) | -0.33 (0.059)
Statistical Analysis 1: Comparison: Pamrevlumab vs Placebo; Test type: Other; p = 0.6579, Mixed Models Analysis; LS Mean Difference = 0.03, 95% CI 2-sided [-0.12 to 0.19], Standard Error of Mean 0.077

2. Secondary Outcome: DB Period: Time to Disease Progression
Description: Time to disease progression was defined as time from randomization to either the first occurrence of an absolute FVC percent predicted (FVCpp) decline of ≥10% from baseline or death, whichever occurred first. 'Median Time to Event' is an estimated value, which was calculated based on Kaplan-Meier method. For an endpoint in which less than half of the participants have encountered the events, the 'Median Time to Event' might be longer than the reported timeframe of 48 weeks.
Time Frame: Up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 184 | 188
weeks | 59.0 [NA to NA] — Due to smaller number of participants with an event, lower and upper limit of 95% confidence interval (CI) could not be calculated. | NA [49.4 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated.

3. Secondary Outcome: DB Period: Change From Baseline in Quantitative Lung Fibrosis (QLF) Volume at Week 48
Description: The QLF volume is calculated as QLF=total lung capacity volume (TLC) * % of quantitative lung fibrosis for fibrosis of the whole lung. LS mean and SE were analyzed using MMRM.
Time Frame: Baseline, Week 48
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: milliliters
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 71 | 76
milliliters | 255.14 (72.028) | 269.15 (60.898)

4. Secondary Outcome: DB Period: Time to First Occurrence of Any Component of the Clinical Composite Endpoint, Whichever Occurred First
Description: The components of the clinical composite endpoints included acute idiopathic pulmonary fibrosis (IPF) exacerbation, respiratory hospitalization, or death. 'Median Time to Event' is an estimated value, which was calculated based on Kaplan-Meier method. For an endpoint in which less than half of the participants have encountered the events, the 'Median Time to Event' might be longer than the reported timeframe of 48 weeks.
Time Frame: Up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 184 | 188
weeks | NA [59.0 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event, median and 95% CI could not be calculated.

5. Secondary Outcome: DB Period: Time to First Acute IPF Exacerbation
Description: 'Median Time to Event' is an estimated value, which was calculated based on Kaplan-Meier method. For an endpoint in which less than half of the participants have encountered the events, the 'Median Time to Event' might be longer than the reported timeframe of 48 weeks.
Time Frame: Up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 184 | 188
weeks | NA [NA to NA] — Due to smaller number of participants with an event, data could not be calculated. | NA [NA to NA] — Due to smaller number of participants with an event, data could not be calculated.

6. Secondary Outcome: DB Period: Time to All-Cause Mortality
Description: as for outcome 5
Time Frame: Up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 184 | 188
weeks | NA [59.0 to NA] — Due to smaller number of participants with an event, median and upper limit of 95% CI could not be calculated. | 62.9 [NA to NA] — Due to smaller number of participants with an event, lower and upper limit of 95% CI could not be calculated.

7. Secondary Outcome: DB Period: Time to First Respiratory Hospitalization
Description: as for outcome 5
Time Frame: Up to Week 48
Population: The ITT population included all randomized participants.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Pamrevlumab | Placebo
Number analyzed (Participants) | 184 | 188
weeks | NA [NA to NA] — Due to smaller number of participants with an event, data could not be calulated. | NA [NA to NA] — Due to smaller number of participants with an event, data could not be calulated.

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to Week 104
Description: As pre-specified, All-cause mortality data were collected and reported for all enrolled participants; and Serious and Non-serious adverse events data were collected and reported for all participants who received any dose of study medication.
Groups:
- DB Period: Pamrevlumab: Participants received pamrevlumab 30 mg/kg, administered by IV infusion, every 3 weeks, for a total of up to 17 infusions over 48 weeks in the DB period.
- DB Period: Placebo: Participants received pamrevlumab-matching placebo, administered by IV infusion every 3 weeks for a total of up to 17 infusions over 48 weeks in the DB period.
- OLE Period: Pamrevlumab: Participants who completed the treatment in DB period and entered in the OLE period, received pamrevlumab 30 mg/kg administered by IV infusion, every 3 weeks for up to 48 weeks.
Arm/Group | DB Period: Pamrevlumab | DB Period: Placebo | OLE Period: Pamrevlumab
All-Cause Mortality (participants affected / at risk) | 16/184 | 15/188 | 12/86
Serious Adverse Events (participants affected / at risk) | 38/183 | 37/188 | 20/86
Other Adverse Events (participants affected / at risk) | 83/183 | 74/188 | 21/86
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Pamrevlumab (N=183) | DB Period: Placebo (N=188) | OLE Period: Pamrevlumab (N=86)
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 0
Acute coronary syndrome (Cardiac disorders) | 0 | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 1
Left ventricular failure (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 0 | 1 | 0
Scleritis (Eye disorders) | 1 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Asthenia (General disorders) | 0 | 1 | 0
Multiple organ dysfunction syndrome (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Sudden death (General disorders) | 0 | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 0 | 0 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0
Empyema (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Nasal abscess (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 9 | 10 | 0
Pneumonia bacterial (Infections and infestations) | 1 | 1 | 0
Pulmonary sepsis (Infections and infestations) | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 1 | 1 | 1
Sepsis (Infections and infestations) | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Clear cell renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0 | 0
Epilepsy (Nervous system disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 0
Parkinson's disease (Nervous system disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 0
Vertebrobasilar stroke (Nervous system disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 1 | 0
Autoimmune nephritis (Renal and urinary disorders) | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 1 | 0
and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 3 | 2 | 2
Chronic respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 9 | 10 | 12
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 2
Peripheral artery aneurysm (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | DB Period: Pamrevlumab (N=183) | DB Period: Placebo (N=188) | OLE Period: Pamrevlumab (N=86)
Diarrhoea (Gastrointestinal disorders) | 14 | 15 | 4
Asthenia (General disorders) | 11 | 7 | 4
Fatigue (General disorders) | 11 | 5 | 0
Bronchitis (Infections and infestations) | 9 | 12 | 0
COVID-19 (Infections and infestations) | 20 | 16 | 8
Nasopharyngitis (Infections and infestations) | 13 | 14 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 26 | 24 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 16 | 12 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The multisite consortium can publish any time after the data is collected and analyzed by FibroGen. The investigator can only publish after the multisite consortium publishes (or tries to publish and fails). FibroGen has 60 days to review a publication and can extend the embargo up to an additional 120 days (or 180 total).

DOCUMENTS (2):
  • Study Protocol (2023-01-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04419558/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-16): https://cdn.clinicaltrials.gov/large-docs/58/NCT04419558/SAP_001.pdf